CLINICAL TRIAL: NCT02570581
Title: MELA Study - Hedonic Study on the Taste of Drugs Crushed in Food: Observational Study Involving 16 Healthy Volunteers
Acronym: MELA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2013-003461-34
Record Dates: First submitted 2015-09-29; First posted 2015-10-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: volonteeres
MeSH Terms: interventions — Gels; Furosemide; Memantine; zopiclone; Alprazolam; Oxazepam; Donepezil; Clopidogrel; Ramipril; Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (24):
- Plain jelly control (Placebo Comparator): Plain jelly control
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Jelly with: Paracetamol (Active Comparator): Jelly with:
  Paracetamol
  Interventions: Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Jelly with Furosemide (Active Comparator): Jelly with Furosemide
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Jelly with Levothyroxine sodium salt (Active Comparator): Jelly with Levothyroxine sodium salt
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Jelly with memantine (Active Comparator): Jelly with memantine
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- jelly with zopiclone (Active Comparator): Jelly with zopiclone
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- jelly with alprazolam (Active Comparator): elly with alprazolam
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- jelly with Oxazepam (Active Comparator): Jelly with Oxazepam
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- jelly with donepezil (Active Comparator): jelly with donepezil
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Jelly with clopidogrel (Active Comparator): jelly with clopidogrel
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- jelly with ramipril (Active Comparator): jelly with ramipril
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- jelly with Paracetamol + Furosemide + Levothyroxine sodium sa (Active Comparator): Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Plain apple compote control (Placebo Comparator): Plain apple compote control
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam
- Apple compote Paracetamol (Active Comparator): Apple compote Paracetamol
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Apple compote Furosemide (Active Comparator): Apple compote Furosemide
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Apple compote Levothyroxine sodium salt (Active Comparator): Apple compote Levothyroxine sodium salt
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Apple compote Memantine (Active Comparator): Apple compote Memantine
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Apple compote Zopiclone (Active Comparator): Apple compote Zopiclone
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Apple compote Alprazolam (Active Comparator): Apple compote Alprazolam
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Apple compote Oxazepam (Active Comparator): Apple compote Oxazepam
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Apple compote Donepezil (Active Comparator): Apple compote Donepezil
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Apple compote Clopidogrel (Active Comparator): Apple compote Clopidogrel
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Ramipril; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Apple compote Ramipril (Active Comparator): Apple compote Ramipril
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain apple compote control
- Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi (Active Comparator): Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopiclone Alprazolam
  Interventions: Other: Jelly with:Paracetamol; Other: Jelly with Furosemide; Other: Jelly with Levothyroxine sodium salt; Other: Jelly with Memantine; Other: Jelly with Zopiclone; Other: Jelly with Alprazolam; Other: Jelly with Oxazepam; Other: Jelly with Donepezil; Other: Jelly with Clopidogrel; Other: Jelly with Ramipril; Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam; Other: Plain jelly control; Other: Apple compote Paracetamol; Other: Apple compote Furosemide; Other: Apple compote Levothyroxine sodium salt; Other: Apple compote Memantine; Other: Apple compote Zopiclone; Other: Apple compote Alprazolam; Other: Apple compote Oxazepam; Other: Apple compote Donepezil; Other: Apple compote Clopidogrel; Other: Apple compote Ramipril; Other: Plain apple compote control

INTERVENTIONS:
Other: Jelly with:Paracetamol — A single dose of each drug will be opened (Paracetamol capsule) or crushed (tablets) in 100 ml of jelly (intervention 1-10) and in 100 ml of apple compote A mix of 6 drugs will be added to 100 ml of jelly (intervention 11) and in 100 ml of apple compote A negative control will consists in 100 ml of plain jelly or apple compote Each participant will receive 24 small transparent plastic glasses ("verrines") randomly allocated from number 1 to number 24, each verrine containing 5 ml of the initial 100 ml drug preparation. The participant will be blind to the verrine content.
  The participant will taste the verrine content with a 1 ml spoon and spit out each spoonful et rinse his or her mouth with plain water (Evian) between two tests.
  The participant will score each verrine numbered 1-24 with a mark ranging from 0 to 10 on the results scoring sheet.
  Unblinding will take place immediately after the end of the test. Every volunteer will propose alternative solutions.
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Jelly with Furosemide
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Jelly with Levothyroxine sodium salt
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Jelly with Memantine
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Jelly with Zopiclone
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril
Other: Jelly with Alprazolam
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Jelly with Oxazepam
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Jelly with Donepezil
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with ramipril; jelly with zopiclone
Other: Jelly with Clopidogrel
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Jelly with Ramipril
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with zopiclone
Other: Jelly with Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Plain jelly control
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Apple compote Paracetamol
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Apple compote Furosemide
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Apple compote Levothyroxine sodium salt
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Apple compote Memantine
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Apple compote Zopiclone
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Apple compote Alprazolam
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Apple compote Oxazepam
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Apple compote Donepezil
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Apple compote Clopidogrel
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Apple compote Ramipril
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Apple compote + Paracetamol + Furosemide + Levothyroxine sodium salt + Memantine + Zopiclone + Alprazolam
  Arms: Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain apple compote control; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone
Other: Plain apple compote control
  Arms: Apple Paracetamol Furosemide Levothyroxine NACL Memantine Zopi; Apple compote Alprazolam; Apple compote Clopidogrel; Apple compote Donepezil; Apple compote Furosemide; Apple compote Levothyroxine sodium salt; Apple compote Memantine; Apple compote Oxazepam; Apple compote Paracetamol; Apple compote Ramipril; Apple compote Zopiclone; Jelly with Furosemide; Jelly with Levothyroxine sodium salt; Jelly with clopidogrel; Jelly with memantine; Jelly with: Paracetamol; Plain jelly control; jelly with Oxazepam; jelly with Paracetamol + Furosemide + Levothyroxine sodium sa; jelly with alprazolam; jelly with donepezil; jelly with ramipril; jelly with zopiclone

SUMMARY:
Elderly people often suffer from chronic pathologies and they are given polypharmacy. In case of swallowing problems, the drugs are crushed and mixed in food, which alters the taste of food and is a cause of anorexia and malnutrition. Gustative side-effects of crushed drugs have nether been investigated. The MELA study is a one session hedonic test involving 16 healthy volunteers. They will score in a blind manner the taste of 10 drugs commonly prescribed in nursing homes, crushed in jelly or apple compote. These volunteers will be 8 food professionals and 8 geriatric care professionals. Thanks to the MELA protocol, they will have a unique opportunity to communicate and propose solutions to this neglected aspect of malnutrition in elderly populations.

DETAILED DESCRIPTION:
Background. Elderly people often suffer from chronic pathologies and they are given polypharmacy. In nursing homes, the residents take an average number of 6 to 8 active principles / day (Reference Geriatrics ward, Nice University Hospital, France), the equivalent of 10 to 20 medicines / day. But 40 % of the residents have swallowing disorders or cognitive impairment: the nursing staff is obliged to crush tablets and capsules and to give them mixed in a compote, a dairy or a jelly, for instance. Some experts groups (OMEDIT) have published a list of drugs authorized to be crushed, because this practice can modify the pharmacokinetics of certain active principles, and render them inactive or even toxic. However, the gustative aspect of crushed drugs has never been investigated.

Main objective. To identify from the advice of healthy volunteers, on the gustative aspect, which medicine it is acceptable or not recommended to add once crushed or opened in food.

Secondary objective. To search for alternative solutions. Type of study. Phase I study on healthy volunteers. It is a cohort study, with a hedonic, descriptive test in a single group and a single one session, to test the taste of 10 drugs crushed in some jelly and apple compote.

Volunteers participating in the study will be 16 healthy volunteers: 8 professionals of the restaurant, the catering, the food aromas, the nutrition and the dietetics, and 8 doctors, pharmacists, dental surgeons, nurses and/or nurse's aides.

Inclusion criteria: healthy volunteers over 18 years, without allergy known about 10 drugs to be tested. Pregnant women will not be included.

Criteria of evaluation:

1. Quantitative: mark from 0 (bad taste) to 10 (no taste or no unpleasant taste) for the jelly and compote specimens mixed with crushed drugs.
2. Qualitative: description of the perceived aroma (acid, bitter, sweet, salty, astringent, pricking, aromatic).

Brief description of the methodology:

The investigator shall test 10 drugs the most prescribed in the Korian group nursing homes, identified as being able to be crushed or opened. The assay will take place during a single one-morning session in a room specifically dedicated to clinical assays and with the help of a nursing staff trained for clinical assays (Nice University Hospital). Medicine will be crushed in parallel in some jelly and apple compote: 10 single drugs, 1 mixture of 6 drugs and 1 comparator (unmodified plain jelly and compote). Every volunteer will make these 24 tests blind and will fill a scoring sheet. He or she will spit out and have an oral rinse with some water between two tests; the dose susceptible to be ingested will be about 1/500th of a unit dosage. Excepted a risk of allergy, the medical risk is thus unimportant for the tasters. Unblinding will take place immediately after the end of the test. Every volunteer will propose alternative solutions.

Individual duration of the study. One morning. Total duration of the study. One year and half, for the organization of the test and the publication of the results.

Expected fallout

* The fight against senile anorexia and malnutrition, in elderly people who are given polypharmacy, by improving care protocols.
* Proposal of alternative solutions such as pediatric or galenic forms if they exist, other food substrates or new additives which would allow to mask the taste of certain drugs crushed in food.
* Incitement in a policy of reduction of drugs for the elderly.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers over 18 years.

Exclusion Criteria:

* pregnant women. Women in age to borne children will perform a urinary test will just before the assay, under the supervision of the Clinical Research Center nurse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Quantitative- compare the taste between specimens | 1 week after the test
  Quantitative: mark from 0 (bad taste) to 10 (no taste or no unpleasant taste) for the jelly and compote specimens added with crushed drugs.

SECONDARY OUTCOMES:
qualitative - description of the perceived aroma | 1 week after the test
  Qualitative: description of the perceived aroma (acid, bitter, sweet, salty, astringent, pricking, aromatic).

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Research - Archet 1 Hospital Nice Hospital, Nice, France